CLINICAL TRIAL: NCT03886974
Title: Transition to Adult Care in Type 1 Diabetes - Understanding Needs, Expectations, and Experiences of Emerging Adults, Parents, and Healthcare Professionals
Brief Title: Transition to Adult Care in Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Sponsor
Other Study IDs: 147-18-DI
Record Dates: First submitted 2019-03-11; First posted 2019-03-22 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Type1diabetes
Keywords: Transition of care; Support networks; Adults with Type 1 diabetes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adults with type 1 diabetes: People with T1D who are 18 years or older.
- Parents of adults with type 1 diabetes: Parents who have adult children with type 1 diabetes.
- Healthcare providers managing patients with type 1 diabetes: Licensed healthcare providers who are managing patients with T1D (whether in adult or pediatric practice).

SUMMARY:
Successful transition to an adult diabetes clinic is an essential part of both clinical and psychosocial care for emerging adults with type 1 diabetes (T1D). Pediatric patients are generally very well supported by their parents, significant others, and multidisciplinary clinical care teams, however, these support networks tend to change once patients reach adulthood and are required to transition to a more independent clinical care model with their adult care providers. This change can often be an overwhelming adjustment with a potential impact on patient's clinical and psychosocial outcomes. As part of the proposed mixed methods study, in Phase 1, the investigators will develop online questionnaires for primary stakeholders in the transition process to improve understanding of their needs, expectations, and experiences around transition. Based on findings from Phase 1, up to 30 individuals from each of the six groups will be interviewed to discuss their responses and better understand their needs around the transition process (Phase 2). Subsequently, findings from the qualitative analyses of the semi-structured interviews will inform the preparation of recommendations that may help facilitate a successful transition for the various stakeholder groups (Phase 3).

DETAILED DESCRIPTION:
The proposed study has been designed to understand needs, expectations, and experiences of emerging adults, parents, and healthcare providers who have or currently are involved in the transition process in T1D. Although, a few previous studies have focused on exploring these aspects of the transition process, these have mostly been at a regional level focusing on a few clinics instead of an attempt to capture responses at a national level. Additionally, as part of this study, each responding stakeholder participant will be requested to invite other other stakeholder group members who they might know to complete the questionnaire (e.g. a T1D patient sharing study information with their parents and their endocrinologist). This would allow the investigators to get a comprehensive picture of the transition process. The study consists of three phases including an online questionnaire (specific to each stakeholder group) (Phase 1), semi-structured phone interviews with a few participants from each stakeholder participant group (Phase 2), and subsequently, developing recommendations for a transition process that aligns the needs and expectations of the various stakeholder groups (Phase 3).

This project has the potential to highlight T1D patients', their families, and providers' concerns and expectations regarding the transition process from a national sample which, could help develop recommendations to implement a patient-centered, successful transition process for emerging adults with T1D.

Specific aims:

Phase 1: To explore needs, expectations, and experiences of emerging adults with T1D, their parents, and healthcare providers around the transition process.

Phase 2: To conduct semi-structured interviews with participants from three stakeholder groups for in-depth understanding of the issues related to the transition process

Phase 3: To develop recommendations for a patient-centered transition process for emerging adults with T1D

ELIGIBILITY:
Inclusion Criteria:

* US residents
* Adults with T1D
* Parents of adults with T1D
* Healthcare providers caring for patients with T1D (in a pediatric or an adult care setting)
* Fluent in the English Language

Exclusion Criteria:

* Adults with T2D

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study surveys will be advertised throughout the USA using various online forums specific to diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Needs assessment for transition of care | Baseline
  Needs assessment questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Harsimran Singh, PhD, Principal Investigator — Mary & Dick Allen Diabetes Center, Hoag Memorial Hospital Presbyterian
Locations (1):
- Mary & Dick Allen Diabetes Center, Hoag Memorial Hospital Presbyterian, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No